CLINICAL TRIAL: NCT01570140
Title: Large Scale Demonstrator, Webportal Diabetes
Acronym: LSD
Status: Completed | Type: Observational
Sponsor: Henk Bilo, MD (Other)
Collaborators: Isala (Other); University Medical Center Groningen (Other)
Responsible Party: Sponsor-Investigator, Henk Bilo, MD, professor, Medical Research Foundation, The Netherlands
Organization: Medical Research Foundation, The Netherlands (Other)
Other Study IDs: LSD
Record Dates: First submitted 2012-03-29; First posted 2012-04-04 (Estimated); Last update posted 2018-03-21 (Actual); Status verified 2018-03

CONDITIONS: Diabetes Mellitus Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Patient Portals

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Web portal users: T2DM patients in the primary care setting, using the web portal.
  Interventions: Behavioral: Web portal

INTERVENTIONS:
Behavioral: Web portal — This study investigates the effects of the voluntarily use of a webportal and its educational content.

SUMMARY:
Rationale: Accounting for the growth, aging and detrimental life style changes in the Dutch population, the investigators expect further growth of number of known diabetes patients. The economic burden with this increase will be enormous, the healthcare system is under increasing pressure to provide better but more time efficient service to more people with limited human resources. the investigators hypothesize that, by increasing the patients self-management by offering remote care services, this reduction of the individual caseload can be achieved.

Objective: Primary objective is to test the hypothesis that the consistent use of a web portal and its educational content and the possibility to review personal diabetes related data for type 2 diabetes patients (T2DM) in the primary care setting, will result in an improvement quality of life.

Study design and methods: In this Prospective observational cohort study the investigators examine the effect of the voluntarily use of a web portal and its educational content. The primary end point is health related quality of life. We predefined a clinically relevant difference of 0.074 in the EQ-5D index score. Secondary endpoints are diabetes-related distress and well being and a selection of clinical measurements, number of contacts with health care provider and the amount of prescribed medication. The participants are being followed for 1-year and the data will be collected at baseline, after 6 months and 12 months.

ELIGIBILITY:
Inclusion Criteria:

* A diagnosis of type 2 diabetes mellitus, as registered in the primary care system under the diagnosis T90.2, and where the GP is defined as the main care giver
* Aged 18 years or older

Exclusion Criteria:

Cohort study:

* None

Intervention study:

* Mental retardation or psychiatric treatment for schizophrenia, organic mental disorder or bipolar disorder currently or in the past
* Insufficient knowledge of the Dutch language to understand the requirements of the study and/or the questions posed in the questionnaires
* Life expectancy < 1 year due to malignancies or other terminal illnesses
* Cognitive impairment, including dementia, that interferes with trial participation
* Any condition that the Investigator and/or Coordinating Investigator feels would interfere with trial participation or evaluation of results

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study consists of people known with type 2 diabetes mellitus who are being guided and treated in primary health care in the Drenthe region of the Netherlands.
Sampling Method: Non-Probability Sample
Enrollment: 350 (Actual)
Dates: Start 2012-05 (Actual); Primary Completion 2015-02 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
Health Related Quality of Life | 12 months
  EQ-5D questionnaire, representing Health Related Quality of Life dimension

SECONDARY OUTCOMES:
Well-being Index: WHO-5 questionnaire | 12 months
  This five items questionnaire covers positive mood, vitality and general interests. The WHO-5 measures not only the absence of symptoms but gives a reliable indication of mental well-being.This includes the following dimensions:
  * Good spirits
  * Relaxation
  * Being Active
  * Waking up fresh and rested
  * Being interested in things
Diabetes-related distress | 12 months
  PAID-5, questionnaire for diabetes-related distress
Assessing self-efficacy | 12 months
  SDSCA, assessing self-efficacy
Evaluation of general practice | 12 months
  Europep questionnaire, evaluation of general practice
Clinical parameters | 12 months
  * Quetelet index (BMI)
  * Systolic/diastolic blood pressure
  * Creatinine
  * Lipid profile fasting
  * Albumin/Creatinine ratio
  * MDRD
  * monofilament test feet
  * SIMMS classification
  * Fundus photo assessment
  * Smoking
  * Use of alcohol
  * FiveShot questionnaire
  * Diabetes medicine
  * Antihypertensiva
  * Antilipaemica
  * Additional medication
  * Cardiovascular complications

CONTACTS AND LOCATIONS:
Locations (1):
- Isala Clinics, Zwolle, Netherlands

REFERENCES:
- [Derived] Mencke R, van der Vaart A, Pasch A, Harms G, Waanders F, Bilo HJG, van Goor H, Hillebrands JL, van Dijk PR. Serum calcification propensity is associated with HbA1c in type 2 diabetes mellitus. BMJ Open Diabetes Res Care. 2021 Feb;9(1):e002016. doi: 10.1136/bmjdrc-2020-002016. PMID 33627317
- [Derived] Waanders F, Dullaart RPF, Vos MJ, Hendriks SH, van Goor H, Bilo HJG, van Dijk PR. Hypomagnesaemia and its determinants in a contemporary primary care cohort of persons with type 2 diabetes. Endocrine. 2020 Jan;67(1):80-86. doi: 10.1007/s12020-019-02116-3. Epub 2019 Oct 24. PMID 31650393
- [Derived] Hendriks SH, Blanker MH, Roelofsen Y, van Hateren KJJ, Groenier KH, Bilo HJG, Kleefstra N. Gender differences in the evaluation of care for patients with type 2 diabetes: a cross-sectional study (ZODIAC-52). BMC Health Serv Res. 2018 Apr 10;18(1):266. doi: 10.1186/s12913-018-3086-x. PMID 29636042
- [Derived] Roelofsen Y, van Vugt M, Hendriks SH, van Hateren KJ, Groenier KH, Snoek FJ, Kleefstra N, Huijsman R, Bilo HJ. Demographical, Clinical, and Psychological Characteristics of Users and Nonusers of an Online Platform for T2DM Patients (e-VitaDM-3/ZODIAC-44). J Diabetes Res. 2016;2016:6343927. doi: 10.1155/2016/6343927. Epub 2015 Nov 22. PMID 26682232
- [Derived] Roelofsen Y, Hendriks SH, Sieverink F, van Vugt M, van Hateren KJ, Snoek FJ, de Wit M, Gans RO, Groenier KH, van Gemert-Pijnen JE, Kleefstra N, Bilo HJ. Design of the e-Vita diabetes mellitus study: effects and use of an interactive online care platform in patients with type 2 diabetes (e-VitaDM-1/ZODIAC-40). BMC Endocr Disord. 2014 Mar 4;14:22. doi: 10.1186/1472-6823-14-22. PMID 24593656